CLINICAL TRIAL: NCT00469937
Title: A Phase I Study of Lithium During Whole Brain Radiotherapy for Patients With Brain Metastases
Brief Title: Ph I Study of Lithium During Whole Brain Radiotherapy For Patients With Brain Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Gius, MD, PhD, Professor; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC RAD 0521; VU-VICC-RAD-0521; VU-IRB-051043
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Neurotoxicity; Solid Tumor
Keywords: radiation toxicity; neurotoxicity; cognitive/functional effects; unspecified adult solid tumor, protocol specific; adult tumors metastatic to brain
MeSH Terms: conditions — Central Nervous System Neoplasms; Neurotoxicity Syndromes; Radiation Injuries; Brain Neoplasms | interventions — Lithium Carbonate; Lithium; Mental Status and Dementia Tests; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Drug: lithium carbonate; Procedure: cognitive assessment; Procedure: quality-of-life assessment; Radiation: radiation therapy

INTERVENTIONS:
Drug: lithium carbonate — Dose levels Neoadjuvant lithium Concurrent lithium Dose level -1 300mg po QD 300mg po QD Dose level (starting dose) 300mg po BID 300mg po BID Dose level 2 300mg po TID 300mg po TID Dose level 3 300mg po QID 300mg po QID
  Other Names: lithium
Procedure: cognitive assessment — cognitive assessment
Procedure: quality-of-life assessment — quality-of-life assessment
Radiation: radiation therapy — Protocol radiotherapy must begin within seven days following initiation of Lithium therapy if day seven falls on a holiday or weekend; it is acceptable to begin treatment the next business day. One treatment of 3Gy will be given daily with the exception of weekends and holidays for a total of (10 fractions) for a total of 30 Gy over 2 to 3 weeks.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs, such as lithium, may protect normal cells from the side effects of radiation therapy. Giving lithium together with radiation therapy may allow a higher dose of radiation therapy to be given so that more tumor cells are killed.

PURPOSE: This phase I trial is studying the side effects and best dose of lithium when given together with whole-brain radiation therapy in treating patients with brain metastases from primary cancer outside the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of concurrent lithium carbonate and whole-brain radiotherapy, as measured by safety and compliance, in patients with primary extracranial malignancy and brain metastases.

OUTLINE: This is an open-label, dose-escalation study of lithium carbonate.

Patients receive oral lithium carbonate twice daily on days 1-7 and 2-4 times daily on days 8-21. Patients undergo whole-brain radiotherapy once daily on days 8-12 and 15-19.

Cohorts of 3-6 patients receive escalating doses of lithium carbonate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Quality of life and mental status are assessed at baseline, on days 1, 8, and 15, at 1-month post-treatment, and then periodically thereafter.

After completion of study treatment, patients are followed at 1 month and then periodically thereafter.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed extracranial primary malignancy

  * Multiple (i.e., > 3) brain metastases OR < 3 metastases with at least 1 metastasis > 4.0 cm in diameter
  * Not eligible for radiosurgery
* No requirement for immediate whole-brain radiotherapy
* No metastases to the midbrain or brainstem

Exclusion Criteria:

* Zubrod performance status 0-2
* Life expectancy ≥ 8 weeks
* Platelet count > 100,000/mm^3
* ANC > 1,500/mm^3
* Hemoglobin ≥ 10 g/dL
* BUN < 25 mg/dL
* Creatinine < 1.5 mg/dL
* Bilirubin < 1.5 mg/dL
* ALT ≤ 2 times normal
* Sodium > 136 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Neurologically stable

  * No seizure disorders or seizures due to brain metastases
* No medical illnesses or psychiatric conditions that would preclude completion of study treatment
* No sensory neuropathy ≥ grade 2
* No bipolar disorder
* No thyroid disease
* No QTc interval prolongation

PRIOR CONCURRENT THERAPY:

* More than 2 weeks since prior and no concurrent chemotherapy
* At least 2 weeks since prior and no concurrent NSAIDs, angiotensin-converting enzyme inhibitors (e.g., enalapril or captopril), calcium channel blockers, diuretics, selective cyclooxygenase-2 inhibitors, acetazolamide, urea, xanthine, or alkalinizing agents (e.g., sodium bicarbonate)
* No prior radiotherapy to the head and neck area
* No prior radiosurgery
* No concurrent radiotherapy to other sites
* No concurrent anticonvulsants due to brain metastases
* No concurrent psychoactive drugs
* No concurrent thyroid medications
* No concurrent amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of concurrent lithium carbonate and whole-brain radiotherapy as measured by safety and compliance | Safety is measured by the rate of grade 3 or worse

CONTACTS AND LOCATIONS:
Overall Officials: Bo Lu, MD, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee